CLINICAL TRIAL: NCT00299572
Title: Can Alendronate Suppress Aortic and Coronary Artery Calcification and Improve Bone Mineral Density in Chronic Peritoneal Dialysis Patients?
Brief Title: Alendronate for Vascular Calcification in Peritoneal Dialysis Patients?
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Far Eastern Memorial Hospital (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 94040
Record Dates: First submitted 2006-03-05; First posted 2006-03-07 (Estimated); Last update posted 2006-03-07 (Estimated); Status verified 2006-03

CONDITIONS: Peritoneal Dialysis
Keywords: alendronate; peritoneal dialysis; vascular calcification; bone mineral density
MeSH Terms: conditions — Vascular Calcification | interventions — Alendronate

INTERVENTIONS:
Drug: alendronate (Fosamax)

SUMMARY:
Hyperphosphatemia is frequently seen in patients with end-stage renal disease (ESRD). Hyperphosphatemia usually results in a high calcium-phosphorus product (CPP) which may subsequently lead to artery and become a risk factor of cardiovascular complications. Alendronate, due to its effect of inhibiting osteoclasts, is approved for treatment of osteoporosis. Previous reports found the use of bisphosphonates could suppress arterial calcification in hemodialysis dialysis patients. The aim of this study is to evaluate the safety and efficacy of alendronate to suppress coronary artery and aortic calcifications, as well as to improve bone density in chronic peritoneal dialysis (PD) patients.

This study will include ESRD patients who had received maintenance PD for more than 3 months, have high CPP level (≧55), and have chest X-ray proven aortic calcification or coronary artery calcification. All participants are randomly allocated to either group 1 or group 2. Group 1 patients receive alendronate 70 mg once weekly in the first 16 weeks, while group 2 patients receive the same dose of drug every week in the second 16 weeks. The extent of coronary artery and aortic calcification is evaluated by using multi-detector spiral computed tomography, whereas bone mineral density is measured by dual-energy X-ray absorptiometry. Both examinations are performed at week 0, 16 and 32 for each participant. Laboratory studies and possible adverse reactions were regularly monitored.

We expect that alendronate can alleviate the progression of arterial calcification or even improve it. Bone density may also be improved after treatment. Besides, we wish to find the independent factor(s) influencing the efficacy of alendronate. These results may help clinical physicians for early intervention and prevention of cardiovascular complications in ESRD patients.

DETAILED DESCRIPTION:
OBJECTIVES The purpose of this study is to determine if long-term use of alendronate can suppress coronary artery and aortic calcification in chronic PD patients. The effect of alendronate on bone mineral density in this patient group is also evaluated.

METHODS

1. Patients To be eligible for the study, patients have to meet all of the following criteria: (1) have received maintenance PD for more than 3 months at Far Eastern Memorial Hospital, (2) have high CPP level (≧55), and (3) have chest X-ray proven aortic calcification or coronary artery calcification proven before. Patients are excluded if they have any one of the following conditions: (1) had been hospitalized in recent 3 months due to severe comorbid diseases, (2) are hypersensitive to alendronate or any of its components, (3) have esophageal diseases (4) are not able to stand or sit upright for 30 minutes, (5) have refractory hypocalcemia, or (6) patients who are pregnant.

   Each eligible participant has to give his/her written informed consent before the start of study. The study should be approved by the Institutional Review Board of the hospital.
2. Study Design The study is a prospective, randomized cross-over study. Fifty patients will be included. All participants are randomly allocated to either group 1 or group 2. Each group consists of 25 patients. Group 1 patients receive alendronate 70 mg once weekly since the first week till the 16th week of the study, while group 2 patients receive the same dose of drug every week since the 17th week till the 32nd week. Group 1 patients will not receive alendronate since the 17th week till the 32nd week, and group 2 patients will not receive alendronate since the first week till the 16 week. The extent of coronary artery and aortic calcification is evaluated by using multi-detector spiral computed tomography, whereas bone mineral density is measured by dual-energy X-ray absorptiometry. Both examinations are performed at week 0, 16 and 32 for each participant. Serum level of calcium should be kept within normal limits and serum level of phosphorus should be kept below 6 mg/dl.

（3）Administration of Alendronate One tablet of alendronate (70 mg per tablet) should be swallowed by each patient once every week with water at least 30 minutes before breakfast, beverage or medication of the day during the treatment period. Patients must not lie down for at least 30 minutes after taking the drug.

（4）Measurement of Coronary Artery and Aortic Calcification Multi-detector spiral computerized tomography (CT) of the chest is performed at week 0, 16 and 32 for each participant to measure the extent of coronary and aortic calcification.

（5）Measurement of Bone Density Dual energy X-ray absorptiometry is performed at week 0, 16 and 32 for each participant to measure the density of bone.

（6）Demographic and Clinical Characteristics of Patients Patients characteristics such as age and sex are documented. Clinical parameters including body height, body weight, duration of dialysis, calcium concentration of dialysate, and medication under use are recorded. Blood pressure is measured at each clinical visit for 3 times after the patient has sit for at least 15 minutes.

（7）Collection of Laboratory Data Fasting serum levels of albumin, phosphorus, calcium, alkaline phosphatase (ALP), intact parathyroid hormone (iPTH) and hemoglobin level of each patient are checked at study entry and once every month. Fasting serum levels of triglyceride, total cholesterol, high-density lipoprotein cholesterol (HDL-chol), low-density lipoprotein cholesterol (LDL-chol), and hypersensitive C-reactive protein (CRP) of each patient are checked at study entry and once every 3 months.

（8）Record of Adverse Effects of Alendronate Any adverse effect of alendronate is recorded every month at clinic visit. （9）Compliance of Patients Compliance of the patients is monitored by using telephone call once every week during the treatment period with alendronate.

（10）Statistical Analysis All values are expressed as mean ± SD. All data are tested for normal distribution before analysis. Differences between mean values of the 2 groups are tested by means of analysis of variance. Group comparisons of categorical variables are analyzed using chi-square test. Multivariate regression is applied to identify independent determinants of coronary artery and aortic calcification. A probability less than 0.05 is considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* receive maintenance peritoneal dialysis for more than 3 months
* have high calcium-phosphate product (>55 (mg/dL)2)
* have chest X-ray proven aortic calcification or coronary artery calcification proven by coronary angiography

Exclusion Criteria:

* had been hospitalized in recent 3 months due to severe comorbid disease
* hypersensitive to alendronate or any of its components
* have esophageal disease
* not able to stand or sit upright for 30 minutes
* have refractory hypocalcemia
* being pregnant

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50
Dates: Start 2006-03; Study Completion 2006-12

PRIMARY OUTCOMES:
1.Changes of calcification score of coronary arteries and aorta
2.Changes of bone density

SECONDARY OUTCOMES:
changes of parathyroid hormone
changes of serum calcium and phosphate level
changes of C reactive protein
changes of lipid profile
adverse reactions

CONTACTS AND LOCATIONS:
Overall Officials: Chun-Fu Lai, M.D., Principal Investigator — Department of Internal Medicine, Far Eastern Memorial Hospital
Locations (1):
- Far Eastern Memorial Hospital, Taipei, Taiwan

REFERENCES:
- [Derived] Hara T, Hijikata Y, Matsubara Y, Watanabe N. Pharmacological interventions versus placebo, no treatment or usual care for osteoporosis in people with chronic kidney disease stages 3-5D. Cochrane Database Syst Rev. 2021 Jul 7;7(7):CD013424. doi: 10.1002/14651858.CD013424.pub2. PMID 34231877